CLINICAL TRIAL: NCT05821751
Title: The Effect of Prebiotic Inulin on Patients Affected by Recurrent/Metastatic Head and Neck Squamous Cell Carcinoma (R/M HNSCC) Treated With Immune Checkpoint Inhibitors (ICIs): Princess Study
Brief Title: The Effect of Prebiotic Inulin on Patients Affected by R/M HNSCC Treated With Immune Checkpoint Inhibitors
Acronym: PRINCESS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione del Piemonte per l'Oncologia (Other)
Collaborators: Ospedale Santa Croce-Carle Cuneo (Other); Università degli Studi di Trento (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CE IRCCS 301/2021
Record Dates: First submitted 2023-01-31; First posted 2023-04-20 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2023-04

CONDITIONS: Head and Neck Squamous Cell Carcinoma
Keywords: microbiome; inulin; Immune Checkpoint Inhibitors; chemotherapy; cytokines; immune cells; HNSCC; Recurrent/Metastatic; Head and Neck Squamous Cell Carcinoma; Carcinoma; Head and Neck Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Neoplasm Metastasis; Carcinoma | interventions — Inulin; pembrolizumab; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): Pembrolizumab in monotherapy or in combination with chemotherapy (platinum + 5 FU) in standard clinical practice according to the international and local guidelines + inulin
  Interventions: Dietary Supplement: inulin; Drug: Pembrolizumab
- Arm B (Experimental): Nivolumab in monotherapy or in combination with chemotherapy (platinum + 5 FU) in standard clinical practice according to the international and local guidelines + inulin
  Interventions: Dietary Supplement: inulin; Drug: Nivolumab

INTERVENTIONS:
Dietary Supplement: inulin — Inulin will be given to enrolled patients according to manufacturer label indications.
  ICIs (i.e. nivolumab and pembrolizumab) alone or in combination with chemotherapy, if clinically indicated, and their administration scheduling will be planned as per international and local guidelines.
Drug: Pembrolizumab — Pembrolizumab in monotherapy or in combination with chemotherapy (platinum + 5 FU) in standard clinical practice according to the international and local guidelines + inulin
  Arms: Arm A
Drug: Nivolumab — Nivolumab in monotherapy or in combination with chemotherapy (platinum + 5 FU) in standard clinical practice according to the international and local guidelines + inulin
  Arms: Arm B

SUMMARY:
The PRINCESS study is a hypothesis-generating, interventional, open-label, non pharmacological trial designed to characterize the translational and clinical implications of the regular assumptions of inulin on Gut Microbiota, circulating cytokines and immune cells dynamics during ICIs +/- chemotherapy on patients affected by R/M HNSCC.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent to study procedures;
2. Male or female, age > 18 years (at the time consent is obtained);
3. Histological or cytological documentation of HNSCC that was diagnosed as recurrent or metastatic and considered incurable by local therapies;
4. Indication to be treated with ICIs monotherapy, either pembrolizumab or nivolumab or in combination with chemotherapy, according to standard clinical practice;
5. ECOG Performance PS score < 2;
6. Adequate kidney, liver and bone marrow function;
7. Will and ability to comply with the protocol.

Exclusion Criteria:

1. Disease that is suitable for local therapy administered with curative intent;
2. Prior therapy with anti-PD-1 or anti-PD-L1 agents;
3. History of severe allergic reactions or hypersensitivity to trial drugs or any of their excipients;
4. Major surgery < 28 days prior to receiving the first dose of study medication;
5. Toxicity from previous anticancer treatment that includes: Grade 3/4 toxicity considered related to prior therapy and that led to treatment discontinuation; toxicity related to prior treatment that has not resolved to > Grade 1;
6. Central nervous system (CNS) metastases and/or carcinomatous meningitis; with the following exception: patients with asymptomatic CNS metastases who are clinically stable and have no requirement for steroids for at least 14 days prior to the first dose of trial treatment. Patients with carcinomatous meningitis or leptomeningeal spread are excluded regardless of clinical stability.
7. Other additional malignancies that are progressing or require active treatment within the last 5 years with the exception of localized basal and squamous cell carcinoma of the skin or cervical cancer in situ.
8. Active autoimmune disease or syndrome that required systemic treatment within the past 2 years (with use of corticosteroids or immunosuppressive drugs). Replacement therapy (thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
9. Systemic steroid therapy (≥10 mg oral prednisone per day or equivalent) or other immunosuppressive agents within 7 days prior to the first dose of trial treatment.
10. Diagnosis of current pneumonitis or history of non-infectious pneumonitis that required steroids or other immunosuppressive agents;
11. Diagnosis of active infection that required systemic antibiotics therapy, orally or intravenous;.
12. Clinically significant cardiovascular disease within the 6 months prior to the first dose of trial treatment with a New York Heart Association (NYHA) grade II or greater congestive heart failure (CHF); symptomatic pericarditis.
13. Known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS) related illness;
14. Any serious and/or unstable medical conditions, psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
15. Receipt of any live vaccine within 30 days of planned start of study therapy.
16. Pregnant, breastfeeding, or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-12-02 (Actual); Primary Completion 2024-12-02 (Estimated); Study Completion 2025-12-02 (Estimated)

PRIMARY OUTCOMES:
Alpha diversity and Beta diversity analysis in the Gut Microbiota | 12 month
  Comparison of gut microbiota diversity with Shannon index in faeces samples. The analyses were conducted using QIIME software
Evaluation of circulating cytokines dynamics | 12 month
  Analysis of multiple cytokines for identify a cytokine signature related to a patient's outcome and be able to recognize patients who will benefit from treatment.
  Plasma Levels of 18 Cytokines TGF-, TNF-, VEGF, INF-, IL-2, IL-4, IL-5, IL-6, IL-8, IL-10, IL-12, IL-13, IL-15, CCL-2, CCL4, CCL-22, and CXCL-10 were evaluated with the Ella Simple Plex system (ProteinSimple™, San Jose, CA, USA)The concentrations were expressed in pg/mL.
  IL-21 was assessed with the ELISA method (R & D System, Minneapolis, MN, USA). The measured optical densities were expressed as pg/mL.
Rate and evaluation of modification of circulating immune-phenotype dynamics | 12 month
  Rate and evaluation of modification of main circulating immune characters as T lymphocytes, B Lymphocytes, Tregs, neutrophils, Natural Killer, NKT, MDSC during study combination treatment
Evaluation of Immune-predictive molecules | 12 month
  Evaluation of immunomodulatory molecules (PD-1; PD-L1/2; HLA- E; TIM3; LAG3; OX40; VISTA; ICOS) will be assessed at each established time point
Overall Survival Rate | through study completion, an average of 1 year
  OS and the correlation with GM diversity and circulating cytokines and immune cells dynamics.

CONTACTS AND LOCATIONS:
Overall Officials: Danilo Galizia, Principal Investigator — FPO IRCCS Candiolo
Locations (1):
- Fondazione del Piemonte per l'Oncologia-IRCCS Candiolo, Candiolo, Turin, Italy

IPD SHARING:
Plan to Share IPD: Yes